CLINICAL TRIAL: NCT00530231
Title: Capsule Endoscopic Miss Rates Determined by Back-to-Back Capsule Endoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Other Study IDs: 2007-05-041
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-05

CONDITIONS: Capsule Endoscopy
Keywords: Capsule endoscopy; Missing rate

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the missing rate of capsule endoscopy using back-to-back capsule endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with obscure gastrointestinal bleeding

Exclusion Criteria:

* Intestinal stenosis or obstruction
* Swallowing difficulty
* History of abdominal surgery
* History of radiation therapy for abdominal or pelvic lesion
* Age < 15 years
* Pregnancy
* Unstable vital sign or massive hematochezia
* Bleeding lesion, mass > 2 cm, or intestinal stenosis found by CT angiography

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Dong Kyung Chang, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea